CLINICAL TRIAL: NCT07139938
Title: Multicenter Study of Spontaneous Correction of Sagittal Imbalance After Isolated Decompression Surgery Without Corrective Fusion Procedure for Lumbar Spinal Stenosis
Brief Title: Spontaneous Correction of Sagittal Imbalance After Isolated Lumbar Decompression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: N.N. Priorov National Medical Research Center of Traumatology and Orthopedics (Other)
Collaborators: Burdenko Neurosurgery Institute (Other); Pirogov National Medical Surgical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS12-05
Record Dates: First submitted 2025-08-15; First posted 2025-08-24 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: LUMBAR STENOSIS; Sagittal Imbalance; Degeneration Lumbar Spine; Lumbar Decompression
Keywords: lumbar stenosis; sagittal imbalance; lumbar decompression
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort (Other): Isolated lumbar decompression
  Interventions: Procedure: Isolated lumbar decomression

INTERVENTIONS:
Procedure: Isolated lumbar decomression — All patients will undergo microsurgical decompression of stenosed neural structures of the lumbar canal at all clinically significant levels with saving the posterior spinal column (type of decompression may be as unilateral, bilateral, or bilateral from a unilateral approach (over-the-top)), including endoscopic decompression.
  Degenerative lumbar stenosis may be caused by thickened yellow and posterior longitudinal ligaments, facet joints hypertrophy, vertebral body osteophytes posteriorly, synovial (facet joints cysts) and disc cysts.

SUMMARY:
Sagittal spinal imbalance may be caused by orthopedic problems, compression of the neural structures of the spinal canal, and pain syndrome (functional imbalance). Sagittal imbalance in combination with appropriate clinical symptoms may require surgical correction of the spine with fixation. However, in some cases, patients experience spontaneous correction of sagittal balance after isolated decompression without any correction or fusion. Therefore, it is necessary to clarify whether isolated decompression may cause spontaneous correction of sagittal imbalance in patients with degenerative lumbar stenosis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 45 and over;
* 2. Radicular leg pain and/or neurogenic claudication with/without back pain, caused by single- or multi-level degenerative lumbar stenosis with/without spodylolisthesis, confirmed by MRI;
* 3. Planned isolated decompression of the spinal canal without implantation of any devices;
* 4. Symptoms persisting for at least 3 months prior to surgery;
* 5. Given written Informed Consent;
* 6. Able and agree to fully comply with the clinical protocol and willing to adhere to follow-up schedule and requirements.

Non-Inclusion Criteria:

* 1. Prior any lumbar surgery;
* 2. Scoliosis of any non-degenerative etiology (due to vertebral fractures, idiopathic, etc.);
* 3. Degenerative scoliosis > 20 degrees;
* 4. Any contraindication or inability to undergo baseline and/or follow up MRI or X-ray as required per protocol;
* 5. Any other condition or situation that the investigator believes may interfere with the safety of the subject or the intent and conduct of the study;

Exclusion Criteria:

* 1. Performed intraoperative discotomy;
* 2. Performed intraoperative iatrogenic instability of the lumbar segment (facetectomy, foraminotomy, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-10-06 (Estimated); Study Completion 2027-10-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in lumbar balance parameters | 3 months postoperatively
  To observe the change from baseline in sagittal vertical axis by full body X-Ray, in mm

SECONDARY OUTCOMES:
Change from baseline in lumbar balance parameters | 12 months postoperatively
  To observe the change from baseline in sagittal vertical axis by full body X-Ray, in mm
Change from baseline in lumbar balance parameters | 3 months and 12 months postoperatively
  To observe the change from baseline in full balance integrated index by full body X-Ray
Change from baseline in lumbar balance parameters | 3 months and 12 months postoperatively
  To observe the change from baseline in lumbar lordosis (L1-S1) by full body X-Ray, in degrees
Change from baseline in lumbar balance parameters | 3 months and 12 months postoperatively
  To observe the change from baseline in low lumbar lordosis (L4-S1) by full body X-Ray, in degrees
Change from baseline in lumbar balance parameters | 3 months and 12 months postoperatively
  To observe the change from baseline in segmental lordosis at operated level by full body X-Ray, in degrees
Change in the cross-sectional area of the dural sac, mm2 | 3 months after surgery
  To observe the change in the cross-sectional area of the dural sac at operated lumbar level by MRI
Change from baseline in Oswestry Disability Index | 3 months and 12 months postoperatively
  To observe the change of Oswestry Disability Index as compared to baseline through follow-up terms (min - 0 - the best result, patient is active; max - 50 - the worst result, patient is not physically active
Change from baseline in Numeric Pain Rating Scale | 2 weeks (or at day of hospital discharge), 3 months, 12 months postoperatively
  To observe the change of Numeric Pain Rating Scale as compared to baseline through follow-up terms (0 - no pain, 10 - unbearable pain)
Change from baseline in Neuropathic Pain 4 Questions | 2 weeks (or at day of hospital discharge), 3 months, 12 months postoperatively
  To observe the change of Neuropathic Pain 4 Questions as compared to baseline through follow-up terms. If the total score is more than 4, the pain is neuropathic.
Change from baseline in The Health Transition Item from SF-36 | 2 weeks (or at day of hospital discharge), 3 months, 12 months postoperatively
  To observe the The Health Transition Item as compared to baseline through follow-up terms (Patient's answers range from 2 - ''Much Better,'' 1 -''Somewhat Better,'' 0 - ''About the Same,'' -1 - ''Somewhat Worse,'' to -2 - ''Much Worse.'')
Change from baseline in posture alignment | 2 weeks (or at day of hospital discharge), 3 months, 12 months postoperatively
  To observe the patient's self-assessment of posture changes as compared to baseline (Patient asked: "How has your posture changed since the surgery?" 1 - better, 0 - unchanged (don't know), -1 - worse
Adverse Events | during study, an average of 12 months
  Document Adverse Events (incl. adverse events related to device) occurrence throughout the study

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Pirogov National Medical Surgical Center, Moscow
  - Burdenko Neurosurgery Institute, Moscow
  - Priorov National Medical Research Center of Traumatology and Orthopedics, Moscow